CLINICAL TRIAL: NCT03470025
Title: Psychological Intervention to Improve the COPD Patients' Psychosocial Well-being
Brief Title: Improving Psychosocial Well-being in COPD Patients in Rehabilitation
Acronym: IMPROVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele Roma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RP 22/17
Record Dates: First submitted 2018-03-06; First posted 2018-03-19 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: COPD
Keywords: Rehabilitation; Psychological Intervention; Quality of life
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Psychosocial Intervention; Nutrition Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Psychological Intervention (Experimental): A weekly combined face to face & telephone-based PI (F-TPI); Psychological Intervention and medical therapy
  Interventions: Other: Psychological Intervention
- A telephone-based PI (TPI) (Experimental): Psychological Intervention - A telephone-based PI (TPI); Psychological Intervention and medical therapy
  Interventions: Other: Psychological Intervention
- Optimal medical therapy (No Intervention): Patients will receive optimal medical therapy

INTERVENTIONS:
Other: Psychological Intervention — 1. F-TPI group will be followed for a period of six months with a telephone-based and a face to face psychological intervention, performed by a clinical psychotherapist .
  2. TPI group will be followed for a period of six months with a TPI characterized by 10 telephone clinical interviews, performed by a clinical psychotherapist.
  3. CTRL group with COPD SoC without PI will follow the standard follow-up program for COPD patients after PR.
  Other Names: Medical therapy
  Arms: A telephone-based PI (TPI); Psychological Intervention

SUMMARY:
Because of a lack of clinical trials, there is currently a paucity of evidence on the most effective strategies to identify and address psychological co-morbidity in COPD, or on targeting these interventions to specific patient groups. The relationship between physiological disease impairment and patient's disease experience is weak. Some patients have highly impaired Quality of life (QoL) despite relatively minor lung function impairment, and others have good QoL despite severe lung function impairment. It is likely that psychological and behavioral factors may be relevant; moreover the coping strategies used by patients and their relationship to individual psychological factors have been incompletely explored. Pulmonary Rehabilitation (PR) is part of integrated COPD patient management and its potential impact on QoL should be underlined: several studies have found that physical exercise has a beneficial effect on depression symptoms [GOLD, 2017].

Before initiating PR a comprehensive and careful assessment should be performed: treatment goals, specific healthcare needs, smoking status, nutritional health, self-management capacity, health educational, psychological health status and social circumstances, medical history and comorbidities, and exercise capabilities and limitations. Moreover, PR has beneficial effects on mood status and daily activities.

Sustaining Pulmonary Rehabilitation benefits and regular exercise over the long term is difficult without any maintenance strategy. The main aim of this study is to assess the Effect of the Psychological Intervention (PI) on Quality of life, psychological status and well-being, and the maintenance of Pulmonary Rehabilitation benefits, in COPD patients.

A PI based on psychoeducation and psychological and emotional support may be a key to improve Quality of life and to bring COPD patients to show a greater awareness of their health status.

DETAILED DESCRIPTION:
In this pilot study we will perform two different methodologies of the Psychological Intervention: a telephone-based Psychological Intervention and combined face to face & telephone-based Psychological Intervention, integrating the COPD rehabilitation.

The study will be carried out in a real life setting. An initial sample of 36 COPD patients satisfying the inclusion criteria and accepting the participation of the study will be enrolled at the PR Unit of the IRCCS "San Raffaele Pisana" Roma-Italy. The study enrollment period will be of maximum six months, the treatment period is of six months, and the interim treatment evaluation is of three months will be performed. Max study duration will be of 12 months.

The participants will be recruited prospectively from consecutively admitted patients to the inpatient PR Unit. Participants will be required to have the diagnosis of COPD according to the ATS' Guideline [Qaseem et al., 2011]. All participants will sign informed consent approved by the Institutional Ethic Committee.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD
* Mini-Mental State Examination (MMSE) ≥ 26
* 6 Minute Walking Test ≥ 90 meters , at admission
* Obtaining Written Informed Consent

Exclusion Criteria:

* Comorbidity influencing respiratory ability and functionality
* Delta 6 Minute Walking Distance < 60 meters, at time of admission

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Health related Quality of Life evaluated by the St. George's Respiratory Questionnaire | day 0 to day 182
  the St. George's Respiratory Questionnaire score
Change in Quality of Life evaluated by the Short Form Health Survey General and Mental Health | day 0 to day 182
  the Short Form Health Survey General and Mental Health score
Change in the degree of enjoyment and satisfaction in areas of daily functioning, evaluated by the Quality Of Life Enjoyment And Satisfaction Questionnaire | day 0 to day 182
  the Quality Of Life Enjoyment And Satisfaction Questionnaire score
Maintenance of Functional Exercise evaluated by the Six Minute Walking Test | day 0 to day 182
  the Six Minute Walking Test score
Maintenance of Respiratory Capacity evaluated by the Borg scale | day 0 to day 182
  the Borg scale score
Assessment of dyspnea in activities of daily living by the Medical Research Council scale | day 0 to day 21 (period of the Pulmonary Rehabilitation )
  the Medical Research Council score
Assessment of Respiratory Capacity by the Maugeri Foundation Respiratory Failure Questionnaire | day 0 to day 21 (period of the Pulmonary Rehabilitation)
  the Maugeri Foundation Respiratory Failure score
Assessment of disability by the Barthel Index | day 0 to day 21 (period of the Pulmonary Rehabilitation )
  Barthel Index score

SECONDARY OUTCOMES:
Change in psychological status evaluated by the Symptom Check List (SCL-90) | day 0 to day 182
  the SCL-90 scores
Assessment of the severity of depression by the Beck Depression Inventory II | day 0 to day 182
  the Beck Depression Inventory score
Assessment of different types of anxiety, state anxiety and trait anxiety, by State-Trait Anxiety Inventory Form Y. | day 0 to day 182
  the State-Trait Anxiety Inventory scores
Change in the use of the Coping Strategies evaluated by Brief-COPE | day 0 to day 182
  Brief-COPE

CONTACTS AND LOCATIONS:
Overall Officials: Giulia Prinzi, MA, Principal Investigator — IRCCS San Raffaele Pisana
Locations (1):
- IRCCS San Raffaele Pisana, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carver CS. You want to measure coping but your protocol's too long: consider the brief COPE. Int J Behav Med. 1997;4(1):92-100. doi: 10.1207/s15327558ijbm0401_6. PMID 16250744
- [Background] Celli B, Tetzlaff K, Criner G, Polkey MI, Sciurba F, Casaburi R, Tal-Singer R, Kawata A, Merrill D, Rennard S; COPD Biomarker Qualification Consortium. The 6-Minute-Walk Distance Test as a Chronic Obstructive Pulmonary Disease Stratification Tool. Insights from the COPD Biomarker Qualification Consortium. Am J Respir Crit Care Med. 2016 Dec 15;194(12):1483-1493. doi: 10.1164/rccm.201508-1653OC. PMID 27332504
- [Background] Chen Q, Wu C, Gao Y, Chen L, Liu Y. A clinical study on the role of psychosomatic therapy in evaluation and treatment of patients with chronic obstructive pulmonary disease complicated with anxiety-depression disorder. Int J Clin Exp Med. 2015 Sep 15;8(9):16613-9. eCollection 2015. PMID 26629192
- [Background] Graydon JE, Ross E. Influence of symptoms, lung function, mood, and social support on level of functioning of patients with COPD. Res Nurs Health. 1995 Dec;18(6):525-33. doi: 10.1002/nur.4770180608. PMID 7480853
- [Background] Guell MR, Cejudo P, Ortega F, Puy MC, Rodriguez-Trigo G, Pijoan JI, Martinez-Indart L, Gorostiza A, Bdeir K, Celli B, Galdiz JB. Benefits of Long-Term Pulmonary Rehabilitation Maintenance Program in Patients with Severe Chronic Obstructive Pulmonary Disease. Three-Year Follow-up. Am J Respir Crit Care Med. 2017 Mar 1;195(5):622-629. doi: 10.1164/rccm.201603-0602OC. PMID 27611807
- [Background] Healy K. A Theory of Human Motivation by Abraham H. Maslow - reflection. Br J Psychiatry. 2016 Apr;208(4):313. doi: 10.1192/bjp.bp.115.179622. No abstract available. PMID 27036694
- [Background] Holland AE, Spruit MA, Troosters T, Puhan MA, Pepin V, Saey D, McCormack MC, Carlin BW, Sciurba FC, Pitta F, Wanger J, MacIntyre N, Kaminsky DA, Culver BH, Revill SM, Hernandes NA, Andrianopoulos V, Camillo CA, Mitchell KE, Lee AL, Hill CJ, Singh SJ. An official European Respiratory Society/American Thoracic Society technical standard: field walking tests in chronic respiratory disease. Eur Respir J. 2014 Dec;44(6):1428-46. doi: 10.1183/09031936.00150314. Epub 2014 Oct 30. PMID 25359355
- [Background] Jones PW, Quirk FH, Baveystock CM, Littlejohns P. A self-complete measure of health status for chronic airflow limitation. The St. George's Respiratory Questionnaire. Am Rev Respir Dis. 1992 Jun;145(6):1321-7. doi: 10.1164/ajrccm/145.6.1321. PMID 1595997
- [Background] Kunik ME, Roundy K, Veazey C, Souchek J, Richardson P, Wray NP, Stanley MA. Surprisingly high prevalence of anxiety and depression in chronic breathing disorders. Chest. 2005 Apr;127(4):1205-11. doi: 10.1378/chest.127.4.1205. PMID 15821196
- [Background] Lazarus RS. Coping theory and research: past, present, and future. Psychosom Med. 1993 May-Jun;55(3):234-47. doi: 10.1097/00006842-199305000-00002. No abstract available. PMID 8346332
- [Background] Martinez FD. Early-Life Origins of Chronic Obstructive Pulmonary Disease. N Engl J Med. 2016 Sep 1;375(9):871-8. doi: 10.1056/NEJMra1603287. No abstract available. PMID 27579637
- [Background] Martinu T, Babyak MA, O'Connell CF, Carney RM, Trulock EP, Davis RD, Blumenthal JA, Palmer SM; INSPIRE Investigators. Baseline 6-min walk distance predicts survival in lung transplant candidates. Am J Transplant. 2008 Jul;8(7):1498-505. doi: 10.1111/j.1600-6143.2008.02264.x. PMID 18510641
- [Background] Maurer J, Rebbapragada V, Borson S, Goldstein R, Kunik ME, Yohannes AM, Hanania NA; ACCP Workshop Panel on Anxiety and Depression in COPD. Anxiety and depression in COPD: current understanding, unanswered questions, and research needs. Chest. 2008 Oct;134(4 Suppl):43S-56S. doi: 10.1378/chest.08-0342. PMID 18842932
- [Background] Perret JL, Walters EH, Abramson MJ, McDonald CF, Dharmage SC. The independent and combined effects of lifetime smoke exposures and asthma as they relate to COPD. Expert Rev Respir Med. 2014 Aug;8(4):503-14. doi: 10.1586/17476348.2014.905913. Epub 2014 May 16. PMID 24834459
- [Background] Qaseem A, Wilt TJ, Weinberger SE, Hanania NA, Criner G, van der Molen T, Marciniuk DD, Denberg T, Schunemann H, Wedzicha W, MacDonald R, Shekelle P; American College of Physicians; American College of Chest Physicians; American Thoracic Society; European Respiratory Society. Diagnosis and management of stable chronic obstructive pulmonary disease: a clinical practice guideline update from the American College of Physicians, American College of Chest Physicians, American Thoracic Society, and European Respiratory Society. Ann Intern Med. 2011 Aug 2;155(3):179-91. doi: 10.7326/0003-4819-155-3-201108020-00008. PMID 21810710
- [Background] Russo P, Prinzi G, Kisialiou A, Cardaci V, Stirpe E, Conti V, Fini M, Bonassi S. WITHDRAWN: Action plans and coping strategies in elderly COPD patients influence the result of pulmonary rehabilitation: an observational study. Eur J Phys Rehabil Med. 2017 Apr 14. doi: 10.23736/S1973-9087.17.04501-4. Online ahead of print. PMID 28417609
- [Background] Smoller JW, Pollack MH, Otto MW, Rosenbaum JF, Kradin RL. Panic anxiety, dyspnea, and respiratory disease. Theoretical and clinical considerations. Am J Respir Crit Care Med. 1996 Jul;154(1):6-17. doi: 10.1164/ajrccm.154.1.8680700.
- [Background] Usmani ZA, Carson KV, Heslop K, Esterman AJ, De Soyza A, Smith BJ. Psychological therapies for the treatment of anxiety disorders in chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2017 Mar 21;3(3):CD010673. doi: 10.1002/14651858.CD010673.pub2. PMID 28322440
- [Background] van Manen JG, Bindels PJ, Dekker FW, IJzermans CJ, van der Zee JS, Schade E. Risk of depression in patients with chronic obstructive pulmonary disease and its determinants. Thorax. 2002 May;57(5):412-6. doi: 10.1136/thorax.57.5.412. PMID 11978917
- [Background] Vanfleteren LEGW, Spruit MA, Wouters EFM, Franssen FME. Management of chronic obstructive pulmonary disease beyond the lungs. Lancet Respir Med. 2016 Nov;4(11):911-924. doi: 10.1016/S2213-2600(16)00097-7. Epub 2016 Jun 2. PMID 27264777
- [Background] Vogele C, von Leupoldt A. Mental disorders in chronic obstructive pulmonary disease (COPD). Respir Med. 2008 May;102(5):764-73. doi: 10.1016/j.rmed.2007.12.006. Epub 2008 Jan 28. PMID 18222685
- [Background] Woodruff PG, Agusti A, Roche N, Singh D, Martinez FJ. Current concepts in targeting chronic obstructive pulmonary disease pharmacotherapy: making progress towards personalised management. Lancet. 2015 May 2;385(9979):1789-1798. doi: 10.1016/S0140-6736(15)60693-6. PMID 25943943